CLINICAL TRIAL: NCT00573326
Title: Low-Dose Oral Imatinib in the Treatment of Scleroderma Pulmonary Involvement: A Phase II Pilot Study
Brief Title: Low-Dose Oral Imatinib for Scleroderma Pulmonary Involvement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Policlinico (Other)
Collaborators: Università Politecnica delle Marche (Other)
Responsible Party: Paolo Fraticelli/MD, Università Politecnica delle Marche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FARM 69J AJ9; EudraCT code:2007-005322-68
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Imatinib 200 mg p.o. once a day for 6 months
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — 200 mg p.o. once a day for 6 months

SUMMARY:
The purpose of this study is to verify effect and tolerability of imatinib on pulmonary and skin fibrosis in patients affected by systemic sclerosis.

DETAILED DESCRIPTION:
Low-dose Oral Imatinib in the Treatment of Scleroderma Pulmonary Involvement: a Phase II pilot study.

Background and rationale

Systemic sclerosis (SSc; scleroderma) is a rare, multisystem connective tissue disease characterised by widespread microvascular lesions and by the increased deposition of matrix components in the skin and internal organs, with varying degrees of severity.

The incidence of scleroderma appears to have increased from 0.6 new cases annually per million in 1947 to 19 new cases annually in 1991 .

The median survival have been calculated to be approximately 60% at 5 years and 50% at 10 years. The U.S. collaborative study reported a 12 years survival of 30% .

Moreover, patients with scleroderma have double standardized incidence ratio (SIR) of developing cancer compared to the general population .

The burden for the National Health System is relevant, with a cost of Euro 2.900 for a five-days hospitalization per patient and an annual indirect cost of Euro 2.066 per patient .

Unfortunately, despite advances in the therapy of single clinical manifestation of scleroderma, no proven disease-modifying interventions exist for patients at this time. Therapy is symptomatic consisting on vasodilators, steroids, anti-secretive agents is not very effective and immunosuppressive therapy consisting mainly in high-dose cyclophosphamide is associated with serious side effects.

Our purpose is to treat scleroderma skin and pulmonary fibrosis using a therapeutic strategy based on pathogenetic mechanisms.

The etiology of the disease is unknown, but abnormal oxidative stress has been implicated in the pathogenesis of scleroderma and linked to fibroblast activation. Platelet-derived growth factor (PDGF) seems to be a stimulator of the production of reactive oxygen species (ROS) which are key cell transducers of fibroblast proliferation and collagen gene expression . In more details, it has been observed that ROS generation is strictly related to Ha-Ras, and growth-factor activated extracellular signal-regulated kinases 1/2 (Ha-Ras, ERK1/2), with the Ha-Ras- ERK1/2-ROS circuitry amplified in scleroderma fibroblasts . In fact, over-expression of Ha-Ras or ERK 1/2 or high ROS levels induce collagen gene transcription and senescence in normal fibroblasts 6. Since platelet-derived growth factor (PDGF) can induce ROS and Ras-ERK1/2 signaling and since IgG derived from scleroderma patients (SSc IgG) react with human fibroblasts , Svegliati and co-workers sought Ha-Ras-ERK1/2 and ROS stimulatory molecules in the serum of scleroderma patients and provided evidence that serum of scleroderma patients contains stimulatory IgG autoantibodies directed to the PDGF receptor (PDGFR) 5. These autoantibodies trigger the PDGFR, which induces ROS via Ha-Ras and ERK 1/2 signaling and is ultimately responsible for fibroblast activation, a distinctive feature of scleroderma 5.

Pulmonary involvement is present in a considerable part of the patients and is characterized by typical interstitial lung disease. Most of the patients present bilateral basal alveolitis evolving to diffuse fibrosis and restrictive respiratory failure. Lung fibrosis or pulmonary hypertension is the main cause of death in systemic sclerosis.

Imatinib mesylate (STI571 or Gleevec) is a specific inhibitor of the fusion protein Bcr-Abl, the causal agent in chronic myelogenous leukaemia. Other targets ATP-binding site of tyrosine kinases are for PDGF, PDGF-receptor, c-Kit, and SCF.

Daniels and coll. investigated the role of TGF-beta-induced fibrosis mediated by activation of the Abelson (Abl) tyrosine kinase, and using a mouse model of bleomycin-induced pulmonary fibrosis, found a significant inhibition of lung fibrosis by imatinib .

Since imatinib mesylate exerts selective, dual inhibition of the transforming growth factor beta (TGFbeta) and platelet-derived growth factor (PDGF) pathways a recent study was undertaken to test the potential use of imatinib mesylate as an antifibrotic drug also for the treatment of dermal fibrosis in systemic sclerosis (SSc). The authors found that imatinib at biologically relevant concentrations has potent antifibrotic effects in vitro and in vivo, without toxic side effects. They conclude that its favorable pharmacokinetics and clinical experience with its use in other diseases, imatinib mesylate is a promising candidate for the treatment of fibrotic diseases such as SSc.

Moreover Platelet-derived growth factor (PDGF) is a potent smooth muscle cell mitogen that may contribute to smooth muscle hyperplasia during the development of chronic pulmonary hypertension and selective PDGF inhibition may provide a novel therapeutic strategy for the treatment of chronic PH. Pulmonary arterial hypertension, a disorder limited to the pulmonary circulation, is characterized by pulmonary vascular obstruction and variable pulmonary vasoconstriction leading to increased pulmonary vascular resistance and death. Pulmonary hypertension is a frequent complication of lung fibrosis in systemic sclerosis, but can also occur without overt fibrotic pulmonary involvement in particular in the limited form of scleroderma. The PDGF receptor antagonist STI571 (imatinib) reversed advanced pulmonary vascular disease in 2 animal models of pulmonary hypertension regardless of the initiating stimulus and it has been used successfully in single patients resistant to conventional therapy .

Actually, is approved for the treatment of chronic myelogenous leukemia 7 and progressed malignant gastrointestinal stromal tumors; since altered PDGF signaling play an important role in the skin and pulmonary fibrosis, Imatinib can have therapeutic potential in the treatment of disorders accompanied by overexpression of this growth factor. Since fibrotic complication are disfiguring and responsible for great suffering and mortality, we expect that this drug can confer substantial benefit in patient with scleroderma.

Objectives of the study

The specific objective of this study is to verify effect and tolerability of a new therapy on pulmonary and skin fibrosis in patients affected by systemic sclerosis. This therapy is based upon recent data regarding the pathogenesis of scleroderma and is intended to interfere with PDGF receptor tyrosine kinase activity which plays a central role in type I collagen gene expression. The proposed action has the following other objectives: 1. strengthening of a national network composed of centres trained in the use of experimental drugs for this disease, with a special focus on the development of uniform criteria for outcome evaluation, enforcement of communication channels, creation of strategic synergies for the future, through ideas, projects and data exchange; 2. training of young investigators; 3. sharing of advanced experimental techniques and 'rare' biological samples to improve knowledge about pathogenesis of scleroderma, avoiding as well costly overlap.

Type of Study

To evaluate the effect of the Imatinib treatment the study will follow a 'Simon's optimal two-stage design'. This is a typical Phase II design, whose aim is to limit the number of subjects who will undergo an ineffective therapy. This design consists in two subsequent enrolment phases.

Ten patients (variable: n1) are entered into the study in the first stage of the trial. Their outcome will be evaluated after six months of experimental therapy. If there will be fewer than 10% of good responses (variable: P0), then accrual will terminate and the drug will be rejected as being of little interest. Otherwise, accrual will continue to a total of 30 patients (variable: n). All patients will undergo the same experimental treatment and outcome evaluation. At the end of the study the drug will be rejected if the observed response rate will be less than 30% (variable: P1) of evaluable patients.

Variables n1, n, P0, P1 have been calculated to provide a design with a probability of 0.05 or less of accepting a drug worse than P0 after the first stage and a probability of 0.2 or less of rejecting a drug better than P1 at the end of the study.

A comparison with historical controls (SSc with lung disease who underwent immunosuppressive treatment) will be also performed.

Seventy-five historical controls are needed to have a probability 80% or higher to reveal a true difference > 20% (favour experimental drug), hypothesizing a good response rate 0.1 or less in the control population (one-sided, alpha=0,05)3.

ELIGIBILITY:
Inclusion Criteria:

* SSc with active pulmonary involvement refractory to conventional immunosuppressive regimen
* Presence of active interstitial alveolitis (presence of grade 2 exertional dyspnea according to Mahler Dyspnea Index AND worsening of lung function tests PLUS interstitial alveolitis assessed by HRCTscan, ground-glass pattern involving at least two lung segments OR dyspnea (as defined above)PLUS Interstitial alveolitis assessed by HRCTscan (AS DEFINED ABOVE) AND neutrophilic or eosinophilic alveolitis detected through broncoalveolar lavage
* Resistance to conventional immunosuppressive treatment (worsening or lack of improvement of lung function tests after cyclophosphamide therapy, conducted for at least three months, with a cumulative dosage > or = 6 g
* Age 18-80 years
* Ability ti give an informed consent
* Use of an acceptable method of birth control; pregnancy will be ruled out before study beginning

Exclusion Criteria:

* Connective tissue diseases other than SSc
* Smoking Habit
* Pregnancy or lactation
* HBV or HCV infection
* Severe anaemia (Hb< or = 8g/dl)
* Hepatic disease (ALT or ALP>1.5 fold above normal levels)
* Moderate or severe renal failure (creatinine clearance<59ml/min)
* Severe heart failure, with ejection fraction < or = 35% measured by echocardiography
* thyroid disease with clinical evidence of hyperthyroidism treated with substitutive therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of the pulmonary interstitial disease, evaluated by spirometry and DLCO, lung HRCTscan, emogasanalysis. | 1 year

SECONDARY OUTCOMES:
Cutaneous Involvement, evaluated by the modified Rodnan skin score; quality of life and patient physical and emotional well being, evaluated by SF-36 score and HAQ | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Armando Gabrielli, MD, Study Chair — Università Politecnica delle Marche
Locations (1):
- Università Politecnica delle Marche, Ancona, Ancona, Italy

REFERENCES:
- [Derived] Fraticelli P, Gabrielli B, Pomponio G, Valentini G, Bosello S, Riboldi P, Gerosa M, Faggioli P, Giacomelli R, Del Papa N, Gerli R, Lunardi C, Bombardieri S, Malorni W, Corvetta A, Moroncini G, Gabrielli A; Imatinib in Scleroderma Italian Study Group. Low-dose oral imatinib in the treatment of systemic sclerosis interstitial lung disease unresponsive to cyclophosphamide: a phase II pilot study. Arthritis Res Ther. 2014 Jul 8;16(4):R144. doi: 10.1186/ar4606. PMID 25007944